CLINICAL TRIAL: NCT07269990
Title: Evaluation of Bone Behavior in Maxillary Post-extractive Sites Treated With Guided Bone Regeneration (G.B.R.) Techniques in Alveolar Socket Preservation (A.S.P.) Procedures With Different Autologous and Heterologous Biomaterials.
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Foggia (Other)
Responsible Party: Principal Investigator, Filiberto Mastrangelo, Clinical Professor, Principal Investigator, University of Foggia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 7-CE-2023
Record Dates: First submitted 2025-11-25; First posted 2025-12-08 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-01

CONDITIONS: Extracting Own Teeth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- compare different types of biomaterials 4 months after application through the use of ASP Group 1 (Active Comparator)
  Interventions: Procedure: compare different types of biomaterials 4 months after application through the use of ASP compare different types of biomaterials 4 months after application through the use of ASP Group 2
- compare different types of biomaterials 4 months after application through the use of ASP Group 2 (Active Comparator)
  Interventions: Procedure: Comparison of different types of biomaterials 4 months after application through the use of ASP
- compare different types of biomaterials 4 months after application through the use of ASP Group 3 (Active Comparator)
  Interventions: Biological: Comparison different types of biomaterials 4 months after application through the use of ASP
- compare different types of biomaterials 4 months after application through the use of ASP Group 4 (Active Comparator)
  Interventions: Procedure: The aim is to compare different types of biomaterials 4 months after application through the use of ASP
- compare different types of biomaterials 4 months after application through the use of ASP Group 5 (Active Comparator)
  Interventions: Procedure: The aim is to compare different types of biomaterials 4 months after application through the use of ASP

INTERVENTIONS:
Procedure: compare different types of biomaterials 4 months after application through the use of ASP compare different types of biomaterials 4 months after application through the use of ASP Group 2 — The aim is to compare different types of biomaterials 4 months after application through the use of ASP in Group 1
  Arms: compare different types of biomaterials 4 months after application through the use of ASP Group 1
Procedure: Comparison of different types of biomaterials 4 months after application through the use of ASP — The aim is to compare different types of biomaterials 4 months after application through the use of ASP in Group 2
  Arms: compare different types of biomaterials 4 months after application through the use of ASP Group 2
Biological: Comparison different types of biomaterials 4 months after application through the use of ASP — The aim is to compare different types of biomaterials 4 months after application through the use of ASP in Group 3
  Arms: compare different types of biomaterials 4 months after application through the use of ASP Group 3
Procedure: The aim is to compare different types of biomaterials 4 months after application through the use of ASP — The aim is to compare different types of biomaterials 4 months after application through the use of ASP in Group 4
  Arms: compare different types of biomaterials 4 months after application through the use of ASP Group 4
Procedure: The aim is to compare different types of biomaterials 4 months after application through the use of ASP — The aim is to compare different types of biomaterials 4 months after application through the use of ASP in Group 5
  Arms: compare different types of biomaterials 4 months after application through the use of ASP Group 5

SUMMARY:
The maxillary bone atrophies from traumatic, pathological events or related to physiological bone loss after tooth extraction, promoting a decrease in bone volume (vertical-horizontal) which has always been a crucial challenge for the clinician in order to obtain adequate rehabilitations prosthetics.

The results of bone loss induced aesthetic and functional difficulties in achieving surgical and prosthetic rehabilitation of the right dental implant.

Bone loss can be restored with autologous bone grafts and in large bone atrophy of the jaws require complex surgical techniques such as vascularized bone transplantation.

As an alternative to the reconstruction of the maxillary tissue, several surgical techniques have been promoted to prevent or minimize bone resorption through market biomaterials with or without the patient's autologous bone.

To reduce or counteract biological bone resorption, surgeons have promoted alveolar cavity preservation procedures (ASP) with autologous or heterologous graft materials.

Recently, several studies have been published to evaluate the use of demineralized dentin material derived from the extracted tooth to obtain new bone in the maxillary post-extraction site.

The aim of the study is to compare different types of biomaterials 4 months after application through the use of the alveolar socket preservation technique.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients.
* Diagnosis of tooth extraction in the upper or lower jaw.
* Preservation procedures necessary to preserve jawbone volume with Guided
* Bone regeneration with autologous or heterologous biomaterials.

Exclusion Criteria:

* Patients with high risk of receiving the intervention (pre-existing medical conditions/comorbidities/possible adverse events).
* Patients with conditions that may interfere with the evaluation or confound the results. (e.g. they are already taking treatments)
* Patients with refusal to participate, inability to provide data, or at high risk of loss to follow-up.
* Patients with neoplastic pathologies.
* Patients with Radio-Chemo therapies.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-07-03 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Comparison of different biomaterials at 4 months to assess the percentage of residual biomaterial remaining in situ and the percentage of newly formed bone in the regenerated area. | 4 months after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- University of Foggia, Foggia, Foggia, Italy

IPD SHARING:
Plan to Share IPD: Undecided